CLINICAL TRIAL: NCT03814655
Title: Evaluation of the Accuracy of Full Digital Workflow for Guided Implant Surgery Using the R2 Gate Software - a Randomized Clinical Trial (RCT)
Brief Title: Evaluation of the Accuracy of Full Digital Workflow for Guided Implant Surgery Using the R2 Gate Software
Acronym: DIGIMPLGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia Dent Srl (Other)
Collaborators: Carol Davila University of Medicine and Pharmacy (Other); MINEC (Unknown)
Responsible Party: Principal Investigator, Corina Marilena Cristache, Senior Lecturer, DMD, PhD, Dr. Habil., Oral and Maxillofacial Surgeon, Project responsable, Concordia Dent Srl
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MINEC 2/2019
Record Dates: First submitted 2019-01-20; First posted 2019-01-24 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Partially Edentulous Maxilla; Partially Edentulous Mandible
Keywords: Dental implants; digital workflow; guided surgery

STUDY DESIGN:
Intervention Model Description: 54 partially edentulous patients filling the inclusion criteria and with signed consent form are expected to be enrolled in this RCT.
  Each patient will be randomly assigned to one of the following protocol for dental implant insertion:
  * Full digital workflow (n=27 patients/sites),
  * Partially digital workflow (n=27 patients/sites).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full digital workflow (Experimental): 1. Intraoral scan of the partially edentulous site, antagonists and occlusion registration. Radiopaque tray customization over the partially edentulous arch.
  2. CBCT with customized radiopaque tray.
  3. Merging files in R2 Gate software and implant planning.
  4. Guided implant insertion with immediate loading, if possible. Megagen dental implants will be inserted.
  5. Digital impression for final screw-retained crown/bridge.
  6. Assessment of accuracy by comparing stl files (planned and postimplant insertion).
  Interventions: Procedure: Full digital workflow
- Partially digital workflow (Active Comparator): 1. Impression of the edentulous arch and antagonist, occlusion registration. Radiopaque tray customization over the edentulous arch.
  2. CBCT with customized radiopaque tray.
  3. Stone models alone, maximum intercuspal position and customized radiopaque tray will be scanned using a desktop scanner.
  4. Merging files (CBCT and model stl) in R2 Gate software and implant planning.
  5. Guided implant insertion with immediate loading, if possible. Megagen dental implants will be inserted.
  6. Classic impression in customized tray with Impregum.
  7. Functional models will be scanned using the same desktop scanner.
  8. Final screw-retained crown/bridge manufacturing.
  9. Assessment of accuracy by comparing stl files (planned and postimplant insertion).
  Interventions: Procedure: Partially digital workflow

INTERVENTIONS:
Procedure: Full digital workflow — Dental implants will be inserted usig a surgical guide performed after prosthetically driven treatment planning. The workflow will be full digital.
  Arms: Full digital workflow
Procedure: Partially digital workflow — Dental implants will be inserted usig a surgical guide performed after prosthetically driven treatment planning. The workflow will be partially digital.
  Arms: Partially digital workflow

SUMMARY:
The primary aim of the present study is to compare the accuracy of a full digital workflow for dental implants insertion to a partially digital workflow, for a limited edentulous space (1 to 3 dental units), in the maxilla or mandible.

DETAILED DESCRIPTION:
Improvements of dental digital technologies are nowadays enabling clinicians to take the digital impressions of the dental arches, therefore avoiding the use of conventional impression materials. Digital impression procedures are claimed to be an approach to improve the accuracy of dental restorations by minimizing the error prone to conventional impression and gypsum model casting, enabling a high degree of standardization. Patients often prefer intraoral scan when compared to the traditional impression. Digital impression is also recommended when patients have remaining teeth that are extremely mobile or misaligned, due to the risk of exfoliation during the conventional impression procedure.

Despite its poor scientific and clinical evidence, the use of digital technologies into the daily practice registers a rapidly growing.

The precision of digital impressions depends on two different parameters: the resolution of the optical scanning system, and the precision of the matching algorithm which may significantly influence the precision of full arch scans. In order to minimize the effect of matching artifacts, only small parts of the dental arch in close vicinity of the teeth are recommended to be scanned.

For prosthetic restoration purpose, several studies regarding the accuracy of digital vs analogue impression have been performed, but none comparing the accuracy of digital vs partially digital workflow for prosthetically driven guided dental implant insertion.

ELIGIBILITY:
Inclusion Criteria:

* Kennedy Class III partially edentulism with 3 or less missing teeth,
* Good general health with no contraindications for implant surgery,
* Acceptance of dental implant treatment,
* Acceptance of 1 or 2 CBCTs.

Exclusion Criteria:

* Limited bone volume with stadial bone graft requirement,
* Limited mouth opening (impossible to use the surgical stent),
* Parkinson disease (impossible to perform an accurate CBCT).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Accuracy of dental implant insertion | 6 weeks
  Accuracy is described, by the International Organization for Standardization (ISO) standard 5725-1, through the use of two parameters: trueness and precision.
  Trueness refers to the deviation between the actual dimension of the measured object and the resulting measurement, while precision indicates how closely repeated the measurements in a set are.

CONTACTS AND LOCATIONS:
Overall Officials: Corina Marilena Cristache, DMD, PhD, Principal Investigator — Carol Davila University of Medicine and Pharmacy
Locations (2):
- Romania (2):
  - Concordia Dent Clinic, Bucharest
  - "Carol Davila"University of Medicine and Pharmacy, Bucharest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seelbach P, Brueckel C, Wostmann B. Accuracy of digital and conventional impression techniques and workflow. Clin Oral Investig. 2013 Sep;17(7):1759-64. doi: 10.1007/s00784-012-0864-4. Epub 2012 Oct 21. PMID 23086333
- [Background] Mehl A, Ender A, Mormann W, Attin T. Accuracy testing of a new intraoral 3D camera. Int J Comput Dent. 2009;12(1):11-28. English, German. PMID 19213357
- [Background] Pinto A, Raffone C. Postextraction computer-guided implant surgery in partially edentate patients with metal restorations: a case report. Oral Implantol (Rome). 2017 Apr 10;10(1):71-77. doi: 10.11138/orl/2017.10.1.071. eCollection 2017 Jan-Mar. PMID 28757938
- [Background] Joda T, Ferrari M, Braegger U. A digital approach for one-step formation of the supra-implant emergence profile with an individualized CAD/CAM healing abutment. J Prosthodont Res. 2016 Jul;60(3):220-3. doi: 10.1016/j.jpor.2016.01.005. Epub 2016 Feb 9. PMID 26868927
- [Background] Cristache CM, Gurbanescu S. Accuracy Evaluation of a Stereolithographic Surgical Template for Dental Implant Insertion Using 3D Superimposition Protocol. Int J Dent. 2017;2017:4292081. doi: 10.1155/2017/4292081. Epub 2017 May 7. PMID 28555157